CLINICAL TRIAL: NCT03512132
Title: Study of High Density Lipoprotein Function in Type 1 Diabetic Patients With Nephropathy
Acronym: DID&NEPHRO
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: DUVILLARD 2017
Record Dates: First submitted 2018-04-11; First posted 2018-04-30 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- control
  Interventions: Biological: Blood samples; Biological: Urine sample
- T1D with normal albumin levels
  Interventions: Biological: Blood samples; Biological: Urine sample
- T1D with macroalbuminuria
  Interventions: Biological: Blood samples; Biological: Urine sample
- T1D with microalbuminuria
  Interventions: Biological: Blood samples; Biological: Urine sample
- T1D with microalbuminuria and statins
  Interventions: Biological: Blood samples; Biological: Urine sample

INTERVENTIONS:
Biological: Blood samples — 5 EDTA tubes of 7ml and 1 dry tube of 7 ml taken on an empty stomach
Biological: Urine sample — Urine sample on an empty stomach

SUMMARY:
A number of arguments suggest that the deterioration in high density lipoproteins (HDL) functioning may worsen with the development of nephropathy during type 1 diabetes (T1D).

The objective of this study will be to investigate to what extent nephropathy in T1D patients in the microalbuminuria and macroalbuminuria stages, compared to T1D patients without nephropathy, is associated with an alteration in HDL functionality and changes in HDL size and composition (lipids with detailed study of phosphates and sphingolipids, main lipoproteins, inflammatory markers).

ELIGIBILITY:
Inclusion Criteria:

INCLUSION CRITERIA GROUP C (CONTROLS) :

* age > 18 years
* a person who has given oral consent
* Non-diabetics
* Fasting plasma glucose < 6.10 mmol/L (1.1 g/L)
* Triglyceridemia < 1.7 mmol/L (1.5 g/l)
* HDL-C concentration > 1.30 mmol/L (for women and 1.03 mmol/L for men)
* Glomerular filtration flow rate > 90 mL/min/1.73m2 (These thresholds correspond to the standard thresholds for these parameters)

INCLUSION CRITERIA GROUP T1D-N (WITH NORMAL ALBUMINURIA) :

* age > 18 years
* a person who has given oral consent
* Diabetic type 1 (based on the patient's clinical history and/or the presence of anti-glutamate decarboxylase autoantibodies and/or plasma C-peptide less than 0.5 ng/l)
* HbA1c between 6 and 9%.
* normal albuminuria (albumin/creatinine ratio < 2.5 mg/mmol in men and < 3.5 in women)
* glomerular filtration rate > 90 mL/min/1.73m2

INCLUSION CRITERIA GROUP T1D-MICRO (WITH MICROALBUMINURIA)

* age > 18 years
* a person who has given oral consent
* Diabetic type 1 (based on the patient's clinical history and/or the presence of anti-glutamate decarboxylase autoantibodies and/or plasma C-peptide less than 0.5 ng/l)
* HbA1c between 6 and 9%.
* Microalbuminuria (albumin/creatinine ratio > 2.5 mg/mmol in men and > 3.5 in women, and < 30 mg/mmol)
* glomerular filtration rate > 90 mL/min/1.73m2

INCLUSION CRITERIA GROUP T1D-MACRO (WITH MACROALBUMINURIA)

* age > 18 years
* a person who has given oral consent
* Diabetic type 1 (based on the patient's clinical history and/or the presence of anti-glutamate decarboxylase autoantibodies and/or plasma C-peptide less than 0.5 ng/l)
* HbA1c between 6 and 9%.
* Macroalbuminuria (albumin/creatinine ratio > 30 mg/mmol)
* glomerular filtration rate > 45 mL/min/1.73m2

Exclusion Criteria:

* Protected adult
* Patient not affiliated to a social security scheme
* Pregnant or breastfeeding woman
* Drugs interfering with lipid metabolism outside insulin for DT1 : hypolipidemic (only for patients included in the DT1-micro group), corticosteroid, estroprogestogens, retinoic acid, antiproteases.
* BMI > 30 kg/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients treated in the Endocrinology, Diabetology or Nephrology departments of the CHU Dijon Bourgogne or in local nephrology or diabetology practices
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-04-24 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Ability to induce cholesterol efflux | inclusion
  amount of cholesterol captured from cells expressed as %.
Nitric oxide synthesis | inclusion
  variation in the presence of HDL compared to the basal state, i.e. in the absence of HDL
Anti-inflammatory effect | inclusion
  variation in the expression of adhesion molecules (VCAM-1 [vascular cell adhesion molecule 1], ICAM-1 [InterCellular Adhesion Molecule 1] and E selectin) under the influence of TNF-alpha [Tumor Necrosis Factor alpha] in the presence of HDL compared to the absence of HDL.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France